CLINICAL TRIAL: NCT03883854
Title: Percentage and Spectrum of Iron Deficiency in Systolic Heart Failure Patients in Assiut University Hospital
Brief Title: Iron Deficiency in Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Nan Saleeb, Principal Investigator, Assiut University
Other Study IDs: fh
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Full history (including dietary history) 2)clinical examination.
  3)Transthoracic echocardiography :
  * Transthoracic echocardiography for measurement of ejection fraction by simpson s method
    4)Complete blood count.
    5)Complete iron profile
  * serum iron
  * serum ferritin
  * total iron binding capacity
  * transferrin saturation (TSAT) Anemia is defined as hemoglobin (Hb)<13g/dl for males and <12 g/dl for females based on world health organization definition (17) Absolute iron deficiency is serum ferritin (100ug/L) Functional iron deficiency is defined as normal serum ferritin (100-300)with low TAST<20%
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 group: Complete iron profile
  * serum iron
  * serum ferritin
  * total iron binding capacity
  * transferrin saturation (TSAT)

SUMMARY:
Heart failure is a common problem with a prevalence of 1-2% in general population and a major cause of mortality,morbidity and impaired quality of life. Anemia is afrequent comorbidity in stable heart failure patients and it increases morbidity in terms of frequent hospital admissions,impaired exercise capacity,poor quality of life ,and increased mortality

DETAILED DESCRIPTION:
Iron deficiency with or without anemia has been commonly associated with heart failure .Although iron deficiency is the commonest nutritional deficiency worldwide ,affecting more than one-third of the population,its association with heart failure with or without anemia is of growing interest .As iron supplementation improves prognosis in patients with heart failure ,iron deficiency is an attractive therapeutic target.

In 2012 ,the European society of cardiology Guidelines for the diagnosis and treatment of acute and chronic heart failure recognized iron deficiency as a comorbidity in heart failure for the first time and recommended diagnosis of iron deficiency based on iron parameters in all patients suspected of having heart failure.

Iron deficiency can be classified as absolute or functional. Absolute iron deficiency reflects depleted body stores caused by poor dietary intake, impaired gastrointestinal absorption,and chronic blood loss.

Functional iron deficiency is thought to be caused by increased hepcidin production and subsequent inhibition of the iron exporter ferroportin ,leading to impaired absorption and utilization of iron.

Chronic heart failure patients are susceptible to both forms iron deficiency

Aetiology of iron deficiency in chronic heart failure:

The aetiology is multifactorial and complex

1. reduced dietary intake
2. chronic blood loss
3. chronic heart failure causes an inflammatory state which leads to increased hepcidin levels and subsequent iron deficiency due to reduced iron absorption and enhanced reticuloendothelial block

ELIGIBILITY:
Inclusion Criteria:

.100 males or females patients above age of 18years of age and clinically diagnosed with systolic heart failure,ejection fraction<50% by echocardiography admitted in Assiut University hospital

Exclusion Criteria:

.Known to be non cardiac condition causing iron deficiency(haemorrhoids,malignancy).

.other conditions causing fluid overload(eg.renal failure on dialysis ). .congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all participants will undergoe
  1. full history(including dietary history)
  2. clinical examination.
  3. transthoracic echocardiography:for measurement of ejection fraction
  4. complete blood count
  5. complete iron profile: serum iron -serum ferritin-total iron binding capacity-transferrin saturation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2020-03-26 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
percentage of iron deficiency in systolic heart failure patients | 1 year
  systolic heart failure is defined as ejection fraction <50% absolute iron deficiency is serum ferritin<100ug/l.Functional iron deficiency is defined as normal serum ferritin(100-300)ug/l with low transferrin saturation<20%

REFERENCES:
- [Result] Cleland JG, Khand A, Clark A. The heart failure epidemic: exactly how big is it? Eur Heart J. 2001 Apr;22(8):623-6. doi: 10.1053/euhj.2000.2493. No abstract available. PMID 11286518